CLINICAL TRIAL: NCT06384079
Title: Study to Assess Duration of Ureteral Rest Prior to Ureteral Reconstruction Surgery
Brief Title: Duration of Ureteral Rest Prior to Ureteral Reconstruction Surgery
Status: Recruiting | Type: Observational
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Ziho Lee, Principal Investigator, Northwestern University
Other Study IDs: STU00219828
Record Dates: First submitted 2024-02-19; First posted 2024-04-25 (Actual); Last update posted 2024-11-26 (Actual); Status verified 2024-11

CONDITIONS: Ureteral Stricture

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Endoscopic Evaluation: Antegrade and retrograde pyelogram will be completed prior to definitive ureteral repair
  Interventions: Procedure: Antegrade and retrograde pyelogram

INTERVENTIONS:
Procedure: Antegrade and retrograde pyelogram — Participation in the study will guarantee that participants will receive this procedure.

SUMMARY:
Our objective is to assess the effect of duration of ureteral rest, defined as time from conversion of ureteral stent to percutaneous nephrostomy, on stricture length prior to ureteral reconstruction surgery.

ELIGIBILITY:
Inclusion Criteria:

* >18 years of age
* Undergoing ureteral reconstruction surgery for ureteral stricture with conversion of an indwelling stent to a percutaneous nephrostomy tube for ureteral rest
* Willing to sign informed consent form
* Able to read and understand informed consent form

Exclusion Criteria:

* <18 years of age
* Inability to provide informed consent
* Members of vulnerable patient populations

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects over 18 years of age undergoing surgery to fix the ureter.
Sampling Method: Non-Probability Sample
Enrollment: 25 (Estimated)
Dates: Start 2024-09-24 (Actual); Primary Completion 2025-11 (Estimated); Study Completion 2030-11 (Estimated)

PRIMARY OUTCOMES:
Ureteral stricture length measured by antegrade or retrograde pyelogram | 2 weeks and 6 weeks post procedure

SECONDARY OUTCOMES:
Ureteral Stricture Quality will be graded as either narrowed or obliterated segment. | 2 weeks and 6 weeks post procedure

CONTACTS AND LOCATIONS:
Locations (1):
- Northwestern University, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol (2023-10-25): https://cdn.clinicaltrials.gov/large-docs/79/NCT06384079/Prot_000.pdf